CLINICAL TRIAL: NCT04632732
Title: Apelin; ACE2 and Biomarkers of Alveolar-capillary Permeability in SARS-cov-2 (COVID-19).
Acronym: APEL-COVID
Status: Completed | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Principal Investigator, Olivier Lesur, Dr, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Other Study IDs: 2021-3862-APEL-COVID
Record Dates: First submitted 2020-11-03; First posted 2020-11-17 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Covid19
Keywords: Covid19; Apelins; ACE2; ras; ARDS; SARS; lung permeability biomarkers; ELABELA; inflammation; kallikrein-kinin
MeSH Terms: conditions — COVID-19; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — 10cc of blood in EDTA tube and 10cc of blood in heparin tube (up to 5 times). Recovered blood plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- COVID+, SARS: patients COVID+ SARS mechanically ventilated and/or needing more than 6L/min of O2-40% FiO2 for a SpO2 equal or above 90% for more than 24hours.
  Interventions: Diagnostic Test: COVID-19 test; Diagnostic Test: Blood sampling
- COVID+, nonSARS: patients COVID+ nonSARS respiratory symptomatic, with or without lung infiltrates, non mechanically ventilated, and needing less than 6L/min O2-40% FiO2 for a SpO2 equal or above 90%. They are hospitalized on floors (pulmonolgy, internal medecine or in intensives cares units).
  Interventions: Diagnostic Test: COVID-19 test; Diagnostic Test: Blood sampling
- COVID-, ARDS: patients are in ARDS according to the Berlin definition and the lung injury is categorized in the direct form (e.g. pneumonia, aspiration).
  Interventions: Diagnostic Test: COVID-19 test; Diagnostic Test: Blood sampling
- COVID-, nonARDS: patients are not in ARDS according to the Berlin definition but are respiratory symptomatic, with or without lung infiltrates and needing less than 6L O2/min-40% FiO2 for a SpO2 equal or above 90%.
  Interventions: Diagnostic Test: COVID-19 test; Diagnostic Test: Blood sampling
- COVID-, control, MV+: patients hospitalized and mechanically ventilated for non-respiratory reasons (post hoc with sex-age matching).
  Interventions: Diagnostic Test: COVID-19 test; Diagnostic Test: Blood sampling
- COVID-, control, MV-: non mechanically ventilated patients hospitalized for non-respiratory reasons (post hoc with sex-age matching).
  Interventions: Diagnostic Test: COVID-19 test; Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: COVID-19 test — Nasal pharyngeal swab
Diagnostic Test: Blood sampling — 20cc of blood will be collected each 7 days during 28 days.

SUMMARY:
Hypothesis: The apelin/APJ system is involved in the protection of the lung affected by the COVID-19 by interacting with the SARS-coV-2 entry door: the Angiotensin I Converting Enzyme 2 (ACE2) and the renin-angiotensin system (ras). Elevated systemic levels of apelins and ACE2 activity are associated to less critical forms of COVID-19 and characterized by less pulmonary hyperpermeability and inflammation.

Goals: Main: In COVID-19+ patients, to establish the basic knowledge of 1) apelins and related systems (ras and degradation enzymes, of which ACE2) pheno-dynamic profile in bloodstream, 2) pulmonary hyperpermeability profile by biomarker's assessment i) comparison of SARS vs. lesser COVID-19 respiratory injury, and with non COVID-19 ARDS and non ARDS acute respiratory condition. Secondary: To set up links between basic and progressive clinical data (data collection system APEL-COVID).

DETAILED DESCRIPTION:
COVID-19 affects patients by it's entry way: the airways and the deep lung. 20 to 30% of symptomatic adult patients which are hospitalised in or out of the intensive care unit exhibit respiratory distress with major oxygenation index alterations. That syndrome is specifically designated severe acute respiratory syndrome coronavirus 2 (SARS-coV-2). SARS-coV-2 develops 2 weeks after the symptoms start, with a recurring fever, progressing dyspnea and a mortality rate of 10 to 50%. In SARS-coV-2: 1) radiological pulmonary infiltrates are more peripheral and 2) dominancy of hyperinflammation (cytokine storm, of which the interleukine-6 IL-6) and hyperpermeability of the alveolar-capillary barrier is observed, 3) in comparison to a traditional (non COVID) ARDS, the hypoxia generated is exceptionally severe and associated to a pulmonary compliance sparsely reduce in more than 70% of cases.

The Angiotensin I Converting Enzyme 2 (ACE2) is a transmembrane carboxypeptidase of the renin-angiotensin system (ras) implicated in cardiovascular homeostasis. ACE2 counter-regulates the proinflammatory hypertensive ACE1/Angiotensin II (Ang II). ACE2 converts Ang II in Ang1-7 to promote vasodilation, anti-inflammation and tissular protection. ACE2 is expressed abundantly in the lung and is the entry door for many virus like the influenza A, coV-1 and -2. A downregulation of ACE2 activity leads to Ang II excess, with a stimulation of the AngI receptor (AT1R) and an increase of pulmonary vascular permeability, negatively impacting the prognosis of the influenza virus H7N9. More than 85% of pulmonary ACE2 is expressed in apical membrane of alveolar epithelial cell type II (AECII) which are located in the lung distal air spaces at the alveolar-capillary barrier interface. This is where the coV-2 set up and induces the SARS (COVID-19+). AECII regulate the alveolar-capillary barrier permeability. Those produce specific proteins (SP-D or surfactant protein D, and CC-16 or Clara Cell protein) which are released in bloodstream when the alveolar-capillary barrier becomes hyperpermeable and are diagnostic and prognostic biological markers.

The apelin/APJ system could be a protective way by interacting with the renin-angiotensin system (ras) and Angiotensin I Converting Enzyme 2 (ACE2). The apelin/APJ system is recognized to protect and optimize cardiovascular functions. The apelins and receptor APJ operate independently of the catecholaminergic system and constitute a counter regulatory response to the vasopressinergic way with an inodilator activity. The apelin/APJ is largely expressed in the lung and is involved in the reduction of pulmonary inflammation. Apelin-13 stabilizes the mitochondrial function, reduces membrane permeability, prevents apoptosis and stimulates AECII proliferation. The apelin/APJ is reactive to hypoxia like in SARS or ARDS with an increase of blood apelins levels. Apelins are substrates for the ras system and kallikrein/kinin which are producing degradation enzymes like ACE2. Despite this, apelins can reverse a decreased activity of ACE2, and regulate the overproduction of Ang II and the AT1R stimulation which lead to an increase pulmonary vascular permeability and lung edema. APJ is also able to inhibit AT1R by trans-allosteric combination. APJ is a co-receptor for the human and simian immunodeficiency virus, and the apelins block their entry. The proximity between ACE2 and APJ on AECII membranes and their internalization/degradation management in term of the apelins isoform lead to the query of their interaction and the link with their pulmonary protective activity.

Hypothesis: The apelin/APJ system is involved in the protection of the lung affected by the COVID-19 by interacting with the SARS-coV-2 entry door: the Angiotensin I Converting Enzyme 2 (ACE2) and the renin-angiotensin system (ras). Elevated systemic levels of apelins and ACE2 activity are associated to less critical forms of COVID-19 and characterized by less pulmonary hyperpermeability and inflammation.

Goals: Main: In COVID-19+ patients, to establish the basic knowledge of 1) apelins and related systems (ras and degradation enzymes, of which ACE2) pheno-dynamic profile in bloodstream, 2) pulmonary hyperpermeability profile by biomarker's assessment i) comparison of SARS vs. lesser COVID-19 respiratory injury, and with non COVID-19 ARDS and non ARDS acute respiratory condition. Secondary: To set up links between basic and progressive clinical data (data collection system APEL-COVID).

Methods: Observational pilot study of a prospective cohort recruiting in the 36 hours after admission adult patients hospitalized for a symptomatic acute respiratory illness. Groups: 1) COVID+, SARS, MV+ (mechanical ventilation) or not, with more than 6L/min-40% FiO2 for a SpO2 more than 90% for more than 24hrs (n=30); 2) COVID+, non SARS, MV-, with less than 6L/min-40% FiO2 for a SpO2 more than 90% for more than 24hrs (n=30); 3) COVID-, ARDS, MV+, with more than 6L/min-40% FiO2 for a SpO2 more than 90% for more than 24hrs (n=30); 4) COVID-, non ARDS, MV-, with less than 6L/min-40% FiO2 for a SpO2 more than 90% for more than 24hrs (n=30). Given the effects of the pressure generated by mechanical ventilation on epithelial biological markers, 2 sub-groups of 10 controls patients hospitalized for non-respiratory reasons will be constituted post hoc with sex-age matching to the above groups. The patients COVID+ non SARS will be respiratory symptomatic, with or without lung infiltrates and needs in O2 less than 6L/min-40% FiO2 for a SpO2 more than 90% and hospitalized on floors of the pulmonology or internal medicine or in the intensives cares units. The ARDS patients will be selected in the direct form (e.g. pneumonia, aspiration) and the oxygenation index parameters established by Berlin definition.

ELIGIBILITY:
Inclusion Criteria:

* For the 4 -non-control- major groups:
* Adults patients hospitalized for symptomatic acute (presumably infectious) respiratory illness
* In the 36 hours after admission.

Exclusion Criteria:

* Patients already hospitalized for more than 36 hours.
* Pediatric patients.
* Asymptomatic patients.
* Non acute respiratory illness patients.
* Primary pulmonary embolism as causative (i.e pulmonary embolism can be concomitant to respiratory symptoms related to SRAS COVID but not without).
* Exacerbated terminal/severe COPD of Pulmonary fibrosis with or without home oxygen.
* Patients with indirect form of ARDS.
* Cystic fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized on floors (pulmonology or in internal medecine) or in intensive care units of the Sherbrooke hospital/CHUS and patients hospitalized in intensive care units of the Angers hospital/CHUA.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Blood apelins-13/12, -17/16, -36 | 28 days
  Measurement by MS/MS of the blood apelins-13/12, -17/16, -36 each 7 days during 28 days.
Blood angiotensin II | 28 days
  Measurement by ELISA of the blood angiotensin II each 7 days during 28 days.
Blood Clara cell protein (CC16) | 28 days
  Measurement by ELISA of the blood CC16 each 7 days during 28 days.
Blood interleukine-6 (IL-6) | 28 days
  Measurement by ELISA of the blood IL-6 each 7 days during 28 days.
Blood surfactant protein D (SP-D) | 28 days
  Measurement by ELISA of the blood SP-D each 7 days during 28 days.
Plasma ACE2 activity measurement by fluorometry | 28 days
  Measurement of the plasma ACE2 activity each 7 days during 28 days.
Plasma lysyl oxidase activity measurement by fluorometry | 28 days
  Measurement of the plasma lysyl oxidase activity each 7 days during 28 days.
Plasma neprilysin activity measurement by fluorometry | 28 days
  Measurement of the plasma neprilysin activity each 7 days during 28 days.

SECONDARY OUTCOMES:
APACHEII | 28 days
  Prognostic score (APACHEII) each day during 28 days.
Oxygenation index | 28 days
  Oxygenation index each day during 28 days.
Mechanical ventilation | 28 days
  Duration of the mechanical ventilation.
Pulmonary compliance (Dynamic, real-time, on ventilator device: Tidal volume / Plateau pressure - PEEP | 28 days
  Measurement of the pulmonary compliance each day during 28 days.
Length of hospital stay | 28 days
  Measurement of the length of hospital stay and/or mortality in-hospital.
SOFA | 28 days
  Prognostic score (SOFA) each day during 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lesur, MD PhD, Principal Investigator — Sherbrooke University
Locations (1):
- Sherbrooke University, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Sun H, Ning R, Tao Y, Yu C, Deng X, Zhao C, Meng S, Tang F, Xu D. Risk Factors for Mortality in 244 Older Adults With COVID-19 in Wuhan, China: A Retrospective Study. J Am Geriatr Soc. 2020 Jun;68(6):E19-E23. doi: 10.1111/jgs.16533. Epub 2020 May 12. PMID 32383809
- [Background] Nikpouraghdam M, Jalali Farahani A, Alishiri G, Heydari S, Ebrahimnia M, Samadinia H, Sepandi M, Jafari NJ, Izadi M, Qazvini A, Dorostkar R, Tat M, Shahriary A, Farnoosh G, Hosseini Zijoud SR, Taghdir M, Alimohamadi Y, Abbaszadeh S, Gouvarchin Ghaleh HE, Bagheri M. Epidemiological characteristics of coronavirus disease 2019 (COVID-19) patients in IRAN: A single center study. J Clin Virol. 2020 Jun;127:104378. doi: 10.1016/j.jcv.2020.104378. Epub 2020 Apr 21. PMID 32353762
- [Background] Zangrillo A, Beretta L, Scandroglio AM, Monti G, Fominskiy E, Colombo S, Morselli F, Belletti A, Silvani P, Crivellari M, Monaco F, Azzolini ML, Reineke R, Nardelli P, Sartorelli M, Votta CD, Ruggeri A, Ciceri F, De Cobelli F, Tresoldi M, Dagna L, Rovere-Querini P, Serpa Neto A, Bellomo R, Landoni G; COVID-BioB Study Group. Characteristics, treatment, outcomes and cause of death of invasively ventilated patients with COVID-19 ARDS in Milan, Italy. Crit Care Resusc. 2020 Apr 23. Online ahead of print. PMID 32353223
- [Background] Gattinoni L, Coppola S, Cressoni M, Busana M, Rossi S, Chiumello D. COVID-19 Does Not Lead to a "Typical" Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2020 May 15;201(10):1299-1300. doi: 10.1164/rccm.202003-0817LE. No abstract available. PMID 32228035
- [Background] Lu W, Zhang S, Chen B, Chen J, Xian J, Lin Y, Shan H, Su ZZ. A Clinical Study of Noninvasive Assessment of Lung Lesions in Patients with Coronavirus Disease-19 (COVID-19) by Bedside Ultrasound. Ultraschall Med. 2020 Jun;41(3):300-307. doi: 10.1055/a-1154-8795. Epub 2020 Apr 15. PMID 32294796
- [Background] Sayiner A, Cinkooglu A, Tasbakan MS, Basoglu OK, Ceylan N, Savas R, Bayraktaroglu S, Ozhan MH. Radiographic examination of the chest and COVID-19. Ann R Coll Surg Engl. 2020 May;102(5):334. doi: 10.1308/rcsann.2020.0099. No abstract available. PMID 32357307
- [Background] Wu J, Pan J, Teng D, Xu X, Feng J, Chen YC. Interpretation of CT signs of 2019 novel coronavirus (COVID-19) pneumonia. Eur Radiol. 2020 Oct;30(10):5455-5462. doi: 10.1007/s00330-020-06915-5. Epub 2020 May 4. PMID 32367422
- [Background] Toniati P, Piva S, Cattalini M, Garrafa E, Regola F, Castelli F, Franceschini F, Airo P, Bazzani C, Beindorf EA, Berlendis M, Bezzi M, Bossini N, Castellano M, Cattaneo S, Cavazzana I, Contessi GB, Crippa M, Delbarba A, De Peri E, Faletti A, Filippini M, Filippini M, Frassi M, Gaggiotti M, Gorla R, Lanspa M, Lorenzotti S, Marino R, Maroldi R, Metra M, Matteelli A, Modina D, Moioli G, Montani G, Muiesan ML, Odolini S, Peli E, Pesenti S, Pezzoli MC, Pirola I, Pozzi A, Proto A, Rasulo FA, Renisi G, Ricci C, Rizzoni D, Romanelli G, Rossi M, Salvetti M, Scolari F, Signorini L, Taglietti M, Tomasoni G, Tomasoni LR, Turla F, Valsecchi A, Zani D, Zuccala F, Zunica F, Foca E, Andreoli L, Latronico N. Tocilizumab for the treatment of severe COVID-19 pneumonia with hyperinflammatory syndrome and acute respiratory failure: A single center study of 100 patients in Brescia, Italy. Autoimmun Rev. 2020 Jul;19(7):102568. doi: 10.1016/j.autrev.2020.102568. Epub 2020 May 3. PMID 32376398
- [Background] van de Veerdonk FL, Netea MG, van Deuren M, van der Meer JW, de Mast Q, Bruggemann RJ, van der Hoeven H. Kallikrein-kinin blockade in patients with COVID-19 to prevent acute respiratory distress syndrome. Elife. 2020 Apr 27;9:e57555. doi: 10.7554/eLife.57555. PMID 32338605
- [Background] Gralinski LE, Bankhead A 3rd, Jeng S, Menachery VD, Proll S, Belisle SE, Matzke M, Webb-Robertson BJ, Luna ML, Shukla AK, Ferris MT, Bolles M, Chang J, Aicher L, Waters KM, Smith RD, Metz TO, Law GL, Katze MG, McWeeney S, Baric RS. Mechanisms of severe acute respiratory syndrome coronavirus-induced acute lung injury. mBio. 2013 Aug 6;4(4):e00271-13. doi: 10.1128/mBio.00271-13. PMID 23919993
- [Background] Herold S, Gabrielli NM, Vadasz I. Novel concepts of acute lung injury and alveolar-capillary barrier dysfunction. Am J Physiol Lung Cell Mol Physiol. 2013 Nov 15;305(10):L665-81. doi: 10.1152/ajplung.00232.2013. Epub 2013 Sep 13. PMID 24039257
- [Background] Keidar S, Kaplan M, Gamliel-Lazarovich A. ACE2 of the heart: From angiotensin I to angiotensin (1-7). Cardiovasc Res. 2007 Feb 1;73(3):463-9. doi: 10.1016/j.cardiores.2006.09.006. Epub 2006 Sep 19. PMID 17049503
- [Background] Gichuhi PM, Isahakia MA. Electron-microscopic localization of baboon acrosomal antigens using antisperm monoclonal antibody. Acta Anat (Basel). 1992;144(2):178-83. doi: 10.1159/000147304. PMID 1514377
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Wevers BA, van der Hoek L. Renin-angiotensin system in human coronavirus pathogenesis. Future Virol. 2010 Mar;5(2):145-161. doi: 10.2217/fvl.10.4. Epub 2010 Mar 1. PMID 32201502
- [Background] Imai Y, Kuba K, Rao S, Huan Y, Guo F, Guan B, Yang P, Sarao R, Wada T, Leong-Poi H, Crackower MA, Fukamizu A, Hui CC, Hein L, Uhlig S, Slutsky AS, Jiang C, Penninger JM. Angiotensin-converting enzyme 2 protects from severe acute lung failure. Nature. 2005 Jul 7;436(7047):112-6. doi: 10.1038/nature03712. PMID 16001071
- [Background] Kuba K, Imai Y, Rao S, Gao H, Guo F, Guan B, Huan Y, Yang P, Zhang Y, Deng W, Bao L, Zhang B, Liu G, Wang Z, Chappell M, Liu Y, Zheng D, Leibbrandt A, Wada T, Slutsky AS, Liu D, Qin C, Jiang C, Penninger JM. A crucial role of angiotensin converting enzyme 2 (ACE2) in SARS coronavirus-induced lung injury. Nat Med. 2005 Aug;11(8):875-9. doi: 10.1038/nm1267. Epub 2005 Jul 10. PMID 16007097
- [Background] Yang P, Gu H, Zhao Z, Wang W, Cao B, Lai C, Yang X, Zhang L, Duan Y, Zhang S, Chen W, Zhen W, Cai M, Penninger JM, Jiang C, Wang X. Angiotensin-converting enzyme 2 (ACE2) mediates influenza H7N9 virus-induced acute lung injury. Sci Rep. 2014 Nov 13;4:7027. doi: 10.1038/srep07027. PMID 25391767
- [Background] Mossel EC, Wang J, Jeffers S, Edeen KE, Wang S, Cosgrove GP, Funk CJ, Manzer R, Miura TA, Pearson LD, Holmes KV, Mason RJ. SARS-CoV replicates in primary human alveolar type II cell cultures but not in type I-like cells. Virology. 2008 Mar 1;372(1):127-35. doi: 10.1016/j.virol.2007.09.045. Epub 2007 Nov 26. PMID 18022664
- [Background] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Background] Lesur O, Arsalane K, Lane D. Lung alveolar epithelial cell migration in vitro: modulators and regulation processes. Am J Physiol. 1996 Mar;270(3 Pt 1):L311-9. doi: 10.1152/ajplung.1996.270.3.L311. PMID 8638722
- [Background] Berthiaume Y, Lesur O, Dagenais A. Treatment of adult respiratory distress syndrome: plea for rescue therapy of the alveolar epithelium. Thorax. 1999 Feb;54(2):150-60. doi: 10.1136/thx.54.2.150. No abstract available. PMID 10325922
- [Background] Ware LB, Matthay MA. The acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1334-49. doi: 10.1056/NEJM200005043421806. No abstract available. PMID 10793167
- [Background] Lesur O, Berthiaume Y, Blaise G, Damas P, Deland E, Guimond JG, Michel RP. Acute respiratory distress syndrome: 30 years later. Can Respir J. 1999 Jan-Feb;6(1):71-86. doi: 10.1155/1999/812476. PMID 10202222
- [Background] Eisner MD, Parsons P, Matthay MA, Ware L, Greene K; Acute Respiratory Distress Syndrome Network. Plasma surfactant protein levels and clinical outcomes in patients with acute lung injury. Thorax. 2003 Nov;58(11):983-8. doi: 10.1136/thorax.58.11.983. PMID 14586055
- [Background] Park J, Pabon M, Choi AMK, Siempos II, Fredenburgh LE, Baron RM, Jeon K, Chung CR, Yang JH, Park CM, Suh GY. Plasma surfactant protein-D as a diagnostic biomarker for acute respiratory distress syndrome: validation in US and Korean cohorts. BMC Pulm Med. 2017 Dec 15;17(1):204. doi: 10.1186/s12890-017-0532-1. PMID 29246207
- [Background] Lesur O, Langevin S, Berthiaume Y, Legare M, Skrobik Y, Bellemare JF, Levy B, Fortier Y, Lauzier F, Bravo G, Nickmilder M, Rousseau E, Bernard A; Critical Care Research Group of the Quebec Respiratory Health Network. Outcome value of Clara cell protein in serum of patients with acute respiratory distress syndrome. Intensive Care Med. 2006 Aug;32(8):1167-74. doi: 10.1007/s00134-006-0235-1. Epub 2006 Jun 23. PMID 16794838
- [Background] Lesur O, Hermans C, Chalifour JF, Picotte J, Levy B, Bernard A, Lane D. Mechanical ventilation-induced pneumoprotein CC-16 vascular transfer in rats: effect of KGF pretreatment. Am J Physiol Lung Cell Mol Physiol. 2003 Feb;284(2):L410-9. doi: 10.1152/ajplung.00384.2001. Epub 2002 Oct 25. PMID 12533314
- [Background] Wosten-van Asperen RM, Lutter R, Specht PA, Moll GN, van Woensel JB, van der Loos CM, van Goor H, Kamilic J, Florquin S, Bos AP. Acute respiratory distress syndrome leads to reduced ratio of ACE/ACE2 activities and is prevented by angiotensin-(1-7) or an angiotensin II receptor antagonist. J Pathol. 2011 Dec;225(4):618-27. doi: 10.1002/path.2987. Epub 2011 Oct 18. PMID 22009550
- [Background] Zhang R, Pan Y, Fanelli V, Wu S, Luo AA, Islam D, Han B, Mao P, Ghazarian M, Zeng W, Spieth PM, Wang D, Khang J, Mo H, Liu X, Uhlig S, Liu M, Laffey J, Slutsky AS, Li Y, Zhang H. Mechanical Stress and the Induction of Lung Fibrosis via the Midkine Signaling Pathway. Am J Respir Crit Care Med. 2015 Aug 1;192(3):315-23. doi: 10.1164/rccm.201412-2326OC. PMID 25945397
- [Background] Marsault E, Llorens-Cortes C, Iturrioz X, Chun HJ, Lesur O, Oudit GY, Auger-Messier M. The apelinergic system: a perspective on challenges and opportunities in cardiovascular and metabolic disorders. Ann N Y Acad Sci. 2019 Nov;1455(1):12-33. doi: 10.1111/nyas.14123. Epub 2019 Jun 25. PMID 31236974
- [Background] Coquerel D, Sainsily X, Dumont L, Sarret P, Marsault E, Auger-Messier M, Lesur O. The apelinergic system as an alternative to catecholamines in low-output septic shock. Crit Care. 2018 Jan 19;22(1):10. doi: 10.1186/s13054-018-1942-z. PMID 29347994
- [Background] Raab WH, Magerl W, Muller H. Changes in dental blood flow following electrical tooth pulp stimulation--influences of capsaicin and guanethidine. Agents Actions. 1988 Dec;25(3-4):237-9. doi: 10.1007/BF01965022. PMID 3218601
- [Background] Berta J, Kenessey I, Dobos J, Tovari J, Klepetko W, Jan Ankersmit H, Hegedus B, Renyi-Vamos F, Varga J, Lorincz Z, Paku S, Ostoros G, Rozsas A, Timar J, Dome B. Apelin expression in human non-small cell lung cancer: role in angiogenesis and prognosis. J Thorac Oncol. 2010 Aug;5(8):1120-9. doi: 10.1097/JTO.0b013e3181e2c1ff. PMID 20581707
- [Background] Zhang H, Chen S, Zeng M, Lin D, Wang Y, Wen X, Xu C, Yang L, Fan X, Gong Y, Zhang H, Kong X. Apelin-13 Administration Protects Against LPS-Induced Acute Lung Injury by Inhibiting NF-kappaB Pathway and NLRP3 Inflammasome Activation. Cell Physiol Biochem. 2018;49(5):1918-1932. doi: 10.1159/000493653. Epub 2018 Sep 20. PMID 30235451
- [Background] Visser YP, Walther FJ, Laghmani el H, Laarse Av, Wagenaar GT. Apelin attenuates hyperoxic lung and heart injury in neonatal rats. Am J Respir Crit Care Med. 2010 Nov 15;182(10):1239-50. doi: 10.1164/rccm.200909-1361OC. Epub 2010 Jul 9. PMID 20622042
- [Background] Zhang L, Li F, Su X, Li Y, Wang Y, Fang R, Guo Y, Jin T, Shan H, Zhao X, Yang R, Shan H, Liang H. Melatonin prevents lung injury by regulating apelin 13 to improve mitochondrial dysfunction. Exp Mol Med. 2019 Jul 4;51(7):1-12. doi: 10.1038/s12276-019-0273-8. PMID 31273199
- [Background] He L, Xu J, Chen L, Li L. Apelin/APJ signaling in hypoxia-related diseases. Clin Chim Acta. 2015 Dec 7;451(Pt B):191-8. doi: 10.1016/j.cca.2015.09.029. Epub 2015 Oct 3. PMID 26436483
- [Background] Andersen CU, Markvardsen LH, Hilberg O, Simonsen U. Pulmonary apelin levels and effects in rats with hypoxic pulmonary hypertension. Respir Med. 2009 Nov;103(11):1663-71. doi: 10.1016/j.rmed.2009.05.011. Epub 2009 Jun 17. PMID 19539454
- [Background] Wang W, McKinnie SM, Farhan M, Paul M, McDonald T, McLean B, Llorens-Cortes C, Hazra S, Murray AG, Vederas JC, Oudit GY. Angiotensin-Converting Enzyme 2 Metabolizes and Partially Inactivates Pyr-Apelin-13 and Apelin-17: Physiological Effects in the Cardiovascular System. Hypertension. 2016 Aug;68(2):365-77. doi: 10.1161/HYPERTENSIONAHA.115.06892. Epub 2016 May 23. PMID 27217402
- [Background] Siddiquee K, Hampton J, McAnally D, May L, Smith L. The apelin receptor inhibits the angiotensin II type 1 receptor via allosteric trans-inhibition. Br J Pharmacol. 2013 Mar;168(5):1104-17. doi: 10.1111/j.1476-5381.2012.02192.x. PMID 22935142
- [Background] Zhou N, Zhang X, Fan X, Argyris E, Fang J, Acheampong E, DuBois GC, Pomerantz RJ. The N-terminal domain of APJ, a CNS-based coreceptor for HIV-1, is essential for its receptor function and coreceptor activity. Virology. 2003 Dec 5;317(1):84-94. doi: 10.1016/j.virol.2003.08.026. PMID 14675627
- [Background] Zou MX, Liu HY, Haraguchi Y, Soda Y, Tatemoto K, Hoshino H. Apelin peptides block the entry of human immunodeficiency virus (HIV). FEBS Lett. 2000 May 4;473(1):15-8. doi: 10.1016/s0014-5793(00)01487-3. PMID 10802050
- [Background] Zhou N, Fang J, Mukhtar M, Acheampong E, Pomerantz RJ. Inhibition of HIV-1 fusion with small interfering RNAs targeting the chemokine coreceptor CXCR4. Gene Ther. 2004 Dec;11(23):1703-12. doi: 10.1038/sj.gt.3302339. PMID 15306840
- [Background] Imai Y, Kuba K, Penninger JM. The discovery of angiotensin-converting enzyme 2 and its role in acute lung injury in mice. Exp Physiol. 2008 May;93(5):543-8. doi: 10.1113/expphysiol.2007.040048. Epub 2008 Apr 10. PMID 18448662
- [Background] Jia H. Pulmonary Angiotensin-Converting Enzyme 2 (ACE2) and Inflammatory Lung Disease. Shock. 2016 Sep;46(3):239-48. doi: 10.1097/SHK.0000000000000633. PMID 27082314
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Derived] Lesur O, Segal ED, Rego K, Mercat A, Asfar P, Chagnon F. Process-Specific Blood Biomarkers and Outcomes in COVID-19 Versus Non-COVID-19 ARDS (APEL-COVID Study): A Prospective, Observational Cohort Study. J Clin Med. 2024 Oct 4;13(19):5919. doi: 10.3390/jcm13195919. PMID 39407979